CLINICAL TRIAL: NCT04813991
Title: Achieving Peri-Operative Pain Control Without Opioids
Brief Title: Pain Control Without Opioids
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment was never initiated and the PI is leaving the institution so the study is closing.
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO2020-0546
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Perioperative Pain
Keywords: Opioid Analgesic; Ibuprofen; Pain control; Acetaminophen; Laparoscopic Cholescystectomy; Laparoscopic Appendectomy
MeSH Terms: conditions — Agnosia | interventions — Ibuprofen; Oxycodone

STUDY DESIGN:
Intervention Model Description: Randomized Double-Blind Intervention Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 - Ibuprofen Breakthrough (Experimental): 600 mg Ibuprofen for breakthrough pain.
  Interventions: Drug: Ibuprofen 600 mg
- Arm 2 - Oxycodone Breakthrough (Active Comparator): 5 mg of Oxycodone for breakthrough pain.
  Interventions: Drug: OxyCODONE 5 Mg Oral Capsule

INTERVENTIONS:
Drug: Ibuprofen 600 mg — Ibuprofen 600 mg for breakthrough pain.
  Arms: Arm 1 - Ibuprofen Breakthrough
Drug: OxyCODONE 5 Mg Oral Capsule — OxyCODONE 5 Mg Oral Capsule for breakthrough pain.
  Arms: Arm 2 - Oxycodone Breakthrough

SUMMARY:
Adequate outpatient pain control after uncomplicated laparoscopic appendectomy or cholecystectomy can be achieved with minimal breakthrough drugs when used in combination with around the clock non-opioid medications.

DETAILED DESCRIPTION:
Death from opioid overdose is now considered a national emergency. Prescribing of narcotics by physicians, particularly in the perioperative period, remains a significant contributor to opioid addiction. There is a critical need to identify post-operative pain control alternatives that eliminate narcotic usage. Without such information, clinicians will continue to rely on opioids to manage their patients' pain. Prior work supports the notion that there is little difference between the effectiveness of non-steroidal anti-inflammatory drugs (NSAIDs) and that of opioid analgesics in controlling pain following surgical procedures. Recent clinical trials have concluded that a combination of centrally and peripherally acting analgesics improves patients' satisfaction and pain control. Clinical investigators have focused upon limiting opioid use rather than on eliminating the administration of narcotics. not surprisingly, there are no established evidenced-based guidelines for postoperative outpatient non-opioid pain control. The majority of U.S. surgeons continue to rely on opioids as the sole outpatient pain regimen, as suggested by a number of current guidelines.

Our observation is that adequate outpatient pain control after uncomplicated laparoscopic appendectomy or cholecystectomy can be achieved with minimal breakthrough drugs when used in combination with around the clock non-opioid medications.

The amount of opioids prescribed at discharge after laparoscopic appendectomies and cholecystectomies is quite variable. An average prescription is for 200-350 Oral Morphine Equivalents (OME) or 26-46 tabs of 5mg oxycodone with the lowest amount reported of 150 OME (20 tabs of 5mg oxy). One of the most conservative guidelines, the Michigan Surgical Quality Collaborative, recommends prescription of 75 OME after laparoscopic cholecystectomy

AIMS AND OBJECTIVES.

1. Characterize the need for breakthrough pain medication in a cohort of post-operative subjects treated utilizing a 3-day pain regimen consisting of ibuprofen and acetaminophen for postoperative outpatient pain control without the use of opioids.
2. Test the non-inferiority of a regimen consisting of ibuprofen when prescribed on as needed basis in controlling breakthrough pain compared with a regimen using oxycodone.

HYPOTHESIS

We predict that a non-opioid regimen can safely control post-operative pain as effectively as management protocols which include narcotics.

At the completion of the proposed research, our expected outcomes are to demonstrate that the ibuprofen/acetaminophen regimen provides adequate pain relief in patients who undergo uncomplicated laparoscopic cholecystectomy and appendectomy.

We also expect to have demonstrated that when breakthrough pain occurs, non-narcotic medications are as effective as opioids. These findings will be relevant to some 10 million surgeries per year in the U.S. where the patients may never need opioid exposure.

STUDY DESIGN/METHOLOGY

In this single-center, randomized, double-blind intervention trial, adult subjects will be enrolled after routine uncomplicated laparoscopic appendectomy or cholecystectomy for the management of outpatient pain. All participants will provide written informed consent.

All subjects will receive two oral analgesic medications (ibuprofen 600mg and acetaminophen 500mg) three times per day with meals, to consume for three days following discharge from the hospital. For breakthrough pain, with a double-blind approach with opaque capsules for the medications, subjects will be randomized to receive five packages of two pills containing either ibuprofen 600mg (Arm 1) or oxycodone 5mg(Arm 2). They will be instructed to consume breakthrough medications no more than twice per day.

The subjects will maintain a pain log and will record their pain intensity prior to meals each day, and also the maximum pain intensity for the given day, using a verbal pain Numerical Rating Scale (NRS) that ranges from 0 to 10.

A research team member will contact each subject daily by phone for seven days and confirm the subject is consuming their medications and collect information regarding pain intensity.

Subjects will be asked the following questions:

* To rate their pain on a scale of 0 to 10 daily, average and maximum.
* To report the # of breakthrough pain medication pills taken that day and how many total remain

If the subject reports a pain score of 8 or greater after taking the both breakthrough medications during a 24 hour period, they will be considered a study failure. Patient will be told to contact their surgeon for follow up. The research coordinator will follow up these subjects to confirm they have spoken to their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-90
* English or Spanish speaking
* Undergoing routine laparoscopic appendectomy or cholecystectomy
* Able to provide Informed Consent

Exclusion Criteria:

* Current use of methadone
* Opioid use within 30 days prior to hospitalization
* Actively taking anti-inflammatory medications
* History of Adverse Reactions to Study Medications
* Pregnancy
* Currently Breastfeeding
* Ongoing treatment for Peptic Ulcer Disease
* Hepatitis, cirrhosis, severe liver dysfunction (elevated MELD score or LFT's > twice the upper limit of normal.)
* Renal dysfunction with a creatinine more than 25% above age normal values.
* Taking any medicine that might interact with one of the study medications such as SSRI's or Tricyclics, anti-psychotics, anti-malaria medications quinidine or halofantrine, Amiodarone or Dronedarone, diphenhydramine, celecoxib, ranitidine, cimetidine, ritanovir, terbinafine, or St John's Wort

The subject will be withdrawn from the study prior to any randomization if the following occurs:

* Conversion from laparoscopic to open procedure
* Subject does not undergo any operation;
* Subject has a complicated hospital course requiring prolonged hospitalization; subject experiences post-operative complications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Breakthrough Pain | 7 Days
  The need for breakthrough pain medication will be characterized by the estimate of the incidence density for starting breakthrough medication. We will examine potential predictors of the need for breakthrough medication using an actuarial approach

SECONDARY OUTCOMES:
Time-weighted average daily pain score over first three days post-discharge. | 3 Days
  The subjects will maintain a pain log and will record their pain intensity prior to meals each day, and also the maximum pain intensity for the given day, using a verbal pain Numerical Rating Scale (NRS) that ranges from 0 to 10. We will use a general linear model (GLM) approach comparing time-weighted average pain scores over 72-hours as the dependent variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gostin LO, Hodge JG Jr, Noe SA. Reframing the Opioid Epidemic as a National Emergency. JAMA. 2017 Oct 24;318(16):1539-1540. doi: 10.1001/jama.2017.13358. No abstract available. PMID 28832871
- [Background] Tan WH, Yu J, Feaman S, McAllister JM, Kahan LG, Quasebarth MA, Blatnik JA, Eagon JC, Awad MM, Brunt LM. Opioid Medication Use in the Surgical Patient: An Assessment of Prescribing Patterns and Use. J Am Coll Surg. 2018 Aug;227(2):203-211. doi: 10.1016/j.jamcollsurg.2018.04.032. Epub 2018 May 7. PMID 29746919
- [Background] Neuman MD, Bateman BT, Wunsch H. Inappropriate opioid prescription after surgery. Lancet. 2019 Apr 13;393(10180):1547-1557. doi: 10.1016/S0140-6736(19)30428-3. PMID 30983590
- [Background] White PF, Joshi GP, Carpenter RL, Fragen RJ. A comparison of oral ketorolac and hydrocodone-acetaminophen for analgesia after ambulatory surgery: arthroscopy versus laparoscopic tubal ligation. Anesth Analg. 1997 Jul;85(1):37-43. doi: 10.1097/00000539-199707000-00007. PMID 9212119
- [Background] Singla N, Pong A, Newman K; MD-10 Study Group. Combination oxycodone 5 mg/ibuprofen 400 mg for the treatment of pain after abdominal or pelvic surgery in women: a randomized, double-blind, placebo- and active-controlled parallel-group study. Clin Ther. 2005 Jan;27(1):45-57. doi: 10.1016/j.clinthera.2005.01.010. PMID 15763605
- [Background] Mitchell A, van Zanten SV, Inglis K, Porter G. A randomized controlled trial comparing acetaminophen plus ibuprofen versus acetaminophen plus codeine plus caffeine after outpatient general surgery. J Am Coll Surg. 2008 Mar;206(3):472-9. doi: 10.1016/j.jamcollsurg.2007.09.006. Epub 2007 Nov 26. PMID 18308218
- [Background] Kroll PB, Meadows L, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen (i.v.-ibuprofen) in the management of postoperative pain following abdominal hysterectomy. Pain Pract. 2011 Jan-Feb;11(1):23-32. doi: 10.1111/j.1533-2500.2010.00402.x. PMID 20642488
- [Background] Ahiskalioglu EO, Ahiskalioglu A, Aydin P, Yayik AM, Temiz A. Effects of single-dose preemptive intravenous ibuprofen on postoperative opioid consumption and acute pain after laparoscopic cholecystectomy. Medicine (Baltimore). 2017 Feb;96(8):e6200. doi: 10.1097/MD.0000000000006200. PMID 28225506
- [Background] Friedman BW, Dym AA, Davitt M, Holden L, Solorzano C, Esses D, Bijur PE, Gallagher EJ. Naproxen With Cyclobenzaprine, Oxycodone/Acetaminophen, or Placebo for Treating Acute Low Back Pain: A Randomized Clinical Trial. JAMA. 2015 Oct 20;314(15):1572-80. doi: 10.1001/jama.2015.13043. PMID 26501533
- [Background] Gupta A, Abubaker H, Demas E, Ahrendtsen L. A Randomized Trial Comparing the Safety and Efficacy of Intravenous Ibuprofen versus Ibuprofen and Acetaminophen in Knee or Hip Arthroplasty. Pain Physician. 2016 Jul;19(6):349-56. PMID 27454264
- [Background] Chang AK, Bijur PE, Esses D, Barnaby DP, Baer J. Effect of a Single Dose of Oral Opioid and Nonopioid Analgesics on Acute Extremity Pain in the Emergency Department: A Randomized Clinical Trial. JAMA. 2017 Nov 7;318(17):1661-1667. doi: 10.1001/jama.2017.16190. PMID 29114833
- [Background] Krebs EE, Gravely A, Nugent S, Jensen AC, DeRonne B, Goldsmith ES, Kroenke K, Bair MJ, Noorbaloochi S. Effect of Opioid vs Nonopioid Medications on Pain-Related Function in Patients With Chronic Back Pain or Hip or Knee Osteoarthritis Pain: The SPACE Randomized Clinical Trial. JAMA. 2018 Mar 6;319(9):872-882. doi: 10.1001/jama.2018.0899. PMID 29509867
- [Background] Thybo KH, Hagi-Pedersen D, Dahl JB, Wetterslev J, Nersesjan M, Jakobsen JC, Pedersen NA, Overgaard S, Schroder HM, Schmidt H, Bjorck JG, Skovmand K, Frederiksen R, Buus-Nielsen M, Sorensen CV, Kruuse LS, Lindholm P, Mathiesen O. Effect of Combination of Paracetamol (Acetaminophen) and Ibuprofen vs Either Alone on Patient-Controlled Morphine Consumption in the First 24 Hours After Total Hip Arthroplasty: The PANSAID Randomized Clinical Trial. JAMA. 2019 Feb 12;321(6):562-571. doi: 10.1001/jama.2018.22039. PMID 30747964
- [Background] Derry S, Derry CJ, Moore RA. Single dose oral ibuprofen plus oxycodone for acute postoperative pain in adults. Cochrane Database Syst Rev. 2013 Jun 26;2013(6):CD010289. doi: 10.1002/14651858.CD010289.pub2. PMID 23801549
- [Background] Cheung CW, Ching Wong SS, Qiu Q, Wang X. Oral Oxycodone for Acute Postoperative Pain: A Review of Clinical Trials. Pain Physician. 2017 Feb;20(2S):SE33-SE52. PMID 28226340
- [Background] Feinberg AE, Chesney TR, Srikandarajah S, Acuna SA, McLeod RS; Best Practice in Surgery Group. Opioid Use After Discharge in Postoperative Patients: A Systematic Review. Ann Surg. 2018 Jun;267(6):1056-1062. doi: 10.1097/SLA.0000000000002591. PMID 29215370
- [Background] Ladha KS, Neuman MD, Broms G, Bethell J, Bateman BT, Wijeysundera DN, Bell M, Hallqvist L, Svensson T, Newcomb CW, Brensinger CM, Gaskins LJ, Wunsch H. Opioid Prescribing After Surgery in the United States, Canada, and Sweden. JAMA Netw Open. 2019 Sep 4;2(9):e1910734. doi: 10.1001/jamanetworkopen.2019.10734. PMID 31483475
- [Background] Hanson KT, Thiels CA, Polites SF, Gazelka HM, Ray-Zack MD, Zielinski MD, Habermann EB. The opioid epidemic in acute care surgery-Characteristics of overprescribing following laparoscopic cholecystectomy. J Trauma Acute Care Surg. 2018 Jul;85(1):62-70. doi: 10.1097/TA.0000000000001834. PMID 29462081
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Michigan OPEN. Opioid Prescribing Recommendations for Opioid-Naive Patients. https://opioidprescribing.info. Published 2018. Accessed September 17, 2019.
- [Background] Sim V, Hawkins S, Gave AA, Bulanov A, Elabbasy F, Khoury L, Panzo M, Sim E, Cohn S. How low can you go: Achieving postoperative outpatient pain control without opioids. J Trauma Acute Care Surg. 2019 Jul;87(1):100-103. doi: 10.1097/TA.0000000000002295. PMID 31259870
- [Background] Ayad S, Babazade R, Elsharkawy H, Nadar V, Lokhande C, Makarova N, Khanna R, Sessler DI, Turan A. Comparison of Transversus Abdominis Plane Infiltration with Liposomal Bupivacaine versus Continuous Epidural Analgesia versus Intravenous Opioid Analgesia. PLoS One. 2016 Apr 15;11(4):e0153675. doi: 10.1371/journal.pone.0153675. eCollection 2016. PMID 27082959
- [Background] Turan A, Atim A, Dalton JE, Keeyapaj W, Chu W, Bernstein E, Fu A, Jae Ho L, Saager L, Sessler DI. Preoperative angiotensin-converting enzyme inhibitor use is not associated with increased postoperative pain and opioid use. Clin J Pain. 2013 Dec;29(12):1050-6. doi: 10.1097/AJP.0b013e318287a258. PMID 24189772